CLINICAL TRIAL: NCT01263873
Title: Examining the Ease of Intubation Using the Parker Flex-Tip® or a Standard Mallinckrodt® Endotracheal When Using the Glidescope®
Brief Title: Examining the Ease of Intubation Using the Parker Flex-Tip® or a Standard Endotracheal Tube
Acronym: ETT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Brian Radesic, CRNA, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 04-10-05
Record Dates: First submitted 2010-12-17; First posted 2010-12-21 (Estimated); Results first posted 2011-12-19 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Larynx
MeSH Terms: conditions — Laryngeal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mallinckrodt (ETT) (Active Comparator): Artifical Airway Device
  Interventions: Device: Mallinckrodt (ETT)
- Parker Flex Tip (ETT) (Experimental): Artifical Airway Device
  Interventions: Device: Parker Flex-Tip (ETT)

INTERVENTIONS:
Device: Mallinckrodt (ETT) — 7.0 millimeter internal diameter for female 8.0 millimeter internal diameter for male
  Arms: Mallinckrodt (ETT)
Device: Parker Flex-Tip (ETT) — 7.0 millimeter internal diameter for female 8.0 millimeter internal diameter for male
  Arms: Parker Flex Tip (ETT)

SUMMARY:
The purpose of the study is to determine if there are differences related to ease of intubation reported by clinicians who use the Parker Flex-Tip® endotracheal tubes(ETT)compared to the standard Mallinckrodt® (ETT). The problem is two (ETTs), the Parker Flex-Tip® and the Mallinckrodt®, are currently available for use in operative suites for intubation, but few studies have compared these devices with each other. Two research questions to be answered in the study are 1. Is there a difference in the ease of intubation when the Parker Flex-Tip® (ETT) is used when compared to the standard Mallinckrodt® (ETT)? and 2. Are there differences in the number of successful intubations when comparing the Parker Flex-Tip® (ETT) and the standard Mallinckrodt® (ETT)? The hypotheses are the use of the Parker Flex-Tip® (ETT) will demonstrate: 1. Fewer seconds to intubate the trachea. 2. Higher self-reported ease of placement scores and 3. Fewer redirections to intubate the trachea. The number of successful intubations is expected to be the same in both arms of the study.

DETAILED DESCRIPTION:
There are not many different types of (ETT)s with different ends or tips. The standard (ETT) by Mallinckrodt® is a disposable polyvinyl chloride plastic tube that has one hooded Murphy tip eye at the end of the tube. The Murphy tip eye is to help with ventilation and air passage if the main end is occluded with mucus or a foreign body. Another type of (ETT) is the Parker Flex-Tip® (ETT), which has a soft flex-tip that is configured to pass easily through the airway anatomy and has two Murphy tip eyes. Currently there are no published data comparing the Parker Flex-Tip® (ETT) with standard Mallinckrodt® (ETT) when the GlideScope® is used. The data are limited concerning the ease of intubation when using the Parker Flex-Tip® (ETT). The study is a two-factor randomized block intervention study design. Subjects assigned to the first group will be intubated using the standard Mallinckrodt® (ETT). The subjects assigned to the second group will be intubated using the Parker Flex-Tip® (ETT). Randomization will be accomplished using the sealed envelope technique. There are six anesthesia providers who will be using ETTs to intubate. A block design will be used to make sure each anesthesia provider receives the same number of patients randomized to the Mallinckrodt and to the Parker Flex-Tip® (ETT)s.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects that are males and non-pregnant females > or equal to 18 years of age that require a general anesthetic with an (ETT).
2. Able to give informed consent (adults, English reading and speaking)

Exclusion Criteria:

1. Any subject on examination with a mallampati III or greater and/or history of difficult intubation.
2. Any subject with an American Society of Anesthesiologist classification greater than 3.
3. Any subject needing rapid sequence induction.
4. Any subject that the anesthesia provider considers the GlideScope® to be contraindicated.
5. Any subject that an anesthesia provider feels for any reason at any time is not appropriate for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Radesic, DNP, CRNA, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals of Cleveland, Cleveland, Ohio, United States

REFERENCES:
- See also: Parker Flex tip endotracheal tube — http://www.parkermedical.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: October, 2010 through January, 2011 in operative room.
Groups:
- Parker Flex Tip Endotracheal Tube: Parker Flex-Tip® which is a disposable polyvinyl chloride (PVC) Endotracheal tube with a flexible, tapered tip that is anatomically designed to the airway structures.
- Mallinckrodt® Endotracheal Tube: Standard PVC Mallinckrodt® tube used throughout the world for intubating the trachea St. Louis, MO 63134.
Period: Overall Study
Arm/Group | Parker Flex Tip Endotracheal Tube | Mallinckrodt® Endotracheal Tube
Started | 30 | 30
Completed | 29 | 29
Not Completed | 1 | 1
Not completed — One provider unable to complete numbers | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parker Flex Tip Endotracheal Tube | Mallinckrodt® Endotracheal Tube | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 20 | 41
  >=65 years | 9 | 10 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (14) | 51 (19) | 53 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 33
  Male | 12 | 15 | 27
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Ease of Intubation, as Measured by Time in Seconds for ETT Insertion
Description: To measure the ease of intubation by time in seconds for ETT insertion. Time was measured in seconds and started when the anesthesia provider asked for the ETT and stopped once the ETT was placed through the glottis. The time was obtained from video recordings during the intubation by the principal investigator (PI).
Time Frame: Participants were followed for the duration of intubation, an average of 10 minutes
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Parker Flex Tip Endotracheal Tube | Mallinckrodt® Endotracheal Tube
Number analyzed (Participants) | 30 | 30
Seconds | 10.8 (7.6) | 12.7 (7.3)

2. Primary Outcome: Ease of Intubation, as Measured by Number of ETT Redirections
Description: To measure the ease of intubation, once the airway structure was visualized with the GlideScope, the number of ETT redirections at the glottis to intubate the trachea was counted by video recordings by the PI.
Time Frame: Participants were followed for the duration of intubation, an average of 10 minutes
Measure: Mean (Standard Deviation); unit: Number of redirections to place ETT
Arm/Group | Parker Flex Tip Endotracheal Tube | Mallinckrodt® Endotracheal Tube
Number analyzed (Participants) | 30 | 30
Number of redirections to place ETT | 0.7 (1.4) | 1.3 (2.8)

3. Primary Outcome: Ease of Intubation, as Measured by an Ease of ETT Insertion Score.
Description: To measure the ease of intubation, an ease of ETT insertion score was obtained by using a 100 millimeter visual analog scale done by the anesthesia provider doing the intubation. The score of 0 millimeters was the easiest intubation and a score of 100 millimeters was the hardest intubation done by that anesthesia provider.
Time Frame: Participants were followed for the duration of intubation, an average of 10 minutes
Measure: Mean (Standard Deviation); unit: Visual Analog Score in millimeters
Arm/Group | Parker Flex Tip Endotracheal Tube | Mallinckrodt® Endotracheal Tube
Number analyzed (Participants) | 30 | 30
Visual Analog Score in millimeters | 12.7 (12.4) | 17.8 (19.9)

ADVERSE EVENTS:
Arm/Group | Parker Flex Tip Endotracheal Tube | Mallinckrodt® Endotracheal Tube
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
Limitations of this study included an un-blinded use of ETTs

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes